CLINICAL TRIAL: NCT02992002
Title: Influence of Fluid Challenge on End-Expiratory Lung Impedance in Mechanically Ventilated Patients Monitored With Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Becher, Dr Tobias Becher, University Hospital Schleswig-Holstein
Other Study IDs: EIT Fluid Challenge
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Failure; Circulatory Failure; Fluid Responsiveness; Fluid Overload
MeSH Terms: conditions — Respiratory Insufficiency; Shock; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fluid Challenge — Infusion of a standardized amount of crystalloid solution (500 ml) to assess fluid responsiveness by means of changes in cardiac output, assessed by transpulmonary thermodilution.

SUMMARY:
The study investigates the influence of a clinically indicated fluid challenge on end-expiratory lung impedance, assessed by electrical impedance tomography (EIT). EIT data will be collected before, during and after infusion of 500 ml of crystalloid solution in mechanically ventilated patients on an operative intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* patients on mechanical ventilation
* clincial decision to monitor regional ventilation with electrical impedance tomography
* clinical indication for fluid challenge
* established cardiac output monitoring with transpulmonary thermodilution

Exclusion Criteria:

* age < 18 years
* open lung injuries
* instable injury of spine or cranium
* thoracic metal implants
* body mass index > 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed population of intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in end-expiratory lung impedance (EELI) | 15-30 minutes
  To assess the effect of fluid challenge on EELI, the change in EELI during the fluid challenge will be measured by electrical impedance tomography and will be compared to the change in EELI during the last 15 minutes before start of the fluid challenge.

SECONDARY OUTCOMES:
Correlation between change in end-expiratory lung impedance and change in intrathoracic blood volume | 15-30 minutes
  We will assess the correlation between the change in end-expiratory lung impedance during infusion of 500 ml of crystalloid solution and the change in intrathoracic blood volume (assessed by transpulmonary thermodilution) during the same time period.
Fluid responsiveness | 15-30 minutes
  We will investigate whether the ratio of cardiac-related impedance changes to ventilation-related impedance changes, measured by EIT at baseline (i.e. before start of fluid challenge), can predict fluid responsiveness, defined as an increase in stroke volume of greater or equal to 15% compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Schleswig Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No